CLINICAL TRIAL: NCT07108374
Title: Transfusion Recommendations Implemented in the PICU (TRIP)
Brief Title: Implementation of Red Blood Cell Transfusion Recommendations in the Pediatric Intensive Care Unit
Acronym: TRIP
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Lucile Packard Children's Hospital (Other); Children's Hospital of Philadelphia (Other); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Katherine M. Steffen, Clinical Associate Professor, School of Medicine, Department of Pediatrics, Division of Pediatric Critical Care Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 70193; HS029298-03 (Other Grant/Funding Number: AHRQ)
Record Dates: First submitted 2025-06-27; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Red Blood Cell Transfusions
Keywords: Red blood cell transfusions; Pediatric critical care medicine; Implementation Science; Clinical Recommendations

STUDY DESIGN:
Intervention Model Description: This study is best characterized as an interventional prospective cohort study. The investigators will deploy 5 implementation strategies intended to increase use of the red blood cell transfusion recommendations in two pediatric intensive care units. While all strategies will all be used, the investigators anticipate that implementation of the Computerized Clinical Decision Support (CCDS) tools will pose the greatest operational challenges in future studies and thus the focus of this study is on the implementation evaluation of these CCDS tools using an implementation framework (RE-AIM) customized for clinical informatics interventions. The investigators will prospectively evaluate the CCDS tools using the RE-AIM framework using a mixed methods approach that includes data collection from the Electronic Health Record (EHR) based on CCDS use, provider surveys, and data from brief, focused provider interviews.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Implementation strategies to increase use of transfusion recommendations — Five implementation strategies will be employed in this study to enhance use of the blood transfusion recommendations. These include 1) building consensus, 2) provider education, 3) identifying and empowering champions ,4) use of computerized clinical decision support tools, and 5) provide quantitative metric-based feedback. Strategies 1-3 will occur prior to initiation of CCDS tools. All patients admitted to the PICU following the date of CCDS tool initiation will be considered to be part of the post-implementation phase. The investigators will collect data from the EHR on CCDS use and conduct provider surveys and interviews following CCDS tool initiation. Surveys and interviews will be both be conducted at 6 and 12 months post-CCDS tool initiation. Process and outcomes measures will be assessed before an after use of the implementation strategies.

SUMMARY:
Evidence demonstrates that the risks of red blood cell transfusions outweigh benefits in many patients who are hospitalized in the pediatric intensive care unit with increased risk of organ dysfunction, infection, delirium, and death. Recommendations have been developed to restrict transfusion in patients who are unlikely to benefit; however, these recommendations have not been consistently adopted into clinical practice. This study examines use of targeted efforts (implementation strategies) to improve implementation of the recommendations, with a goal of reducing unnecessary transfusions and improving patient outcomes in critically ill children.

ELIGIBILITY:
Inclusion Criteria:

* Employed at Lucile Packard Children's Hospital at Stanford University or the Children's Hospital of Philadelphia AND
* Employed in one of the following roles:
* PICU nurse
* PICU attending
* PICU fellow
* PICU resident
* PICU advanced practice provider
* Other physician or surgeon in subspecialties whose patients regularly receive transfusions in the PICU
* PICU TRIP implementation team member
* PICU nursing leader
* PICU physician leader
* Bood bank leader.

Exclusion Criteria:

* Unwilling to participate
* Directly report to the primary investigator.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-11-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in transfusion recommendation adherence at 18 months (evidence-based threshold alert) | 18 months
  The investigators will assess the mean rate of nonadherent transfusions at monthly intervals in the pre- (12 months prior to CCDS tool initiation) and post-implementation period (18 months following CCDS tool initiation).

SECONDARY OUTCOMES:
Mean change from baseline in transfusion recommendation adherence at 18 months (transfusions that require clinical judgement) | 18 months
  The investigators will assess the mean rate of nonadherent transfusions at monthly intervals in the pre- (12 months prior to CCDS tool initiation) and post-implementation period (18 months following CCDS tool initiation) for transfusions that require provider clinical judgement. Data analysis will be exploratory.
Reach of computerized clinical decision support (CCDS) tools | 18 months
  We will assess Reach of the CCDS tools by assessing the number of triggered CCDS alerts as compared with the total number of patients at risk for unnecessary transfusion (as determined through the PEDSnet database under IRB 16-012878, PEDSnet Master Secondary Use Protocol, under amendment 96, Appendix 28).

OTHER OUTCOMES:
Unintended consequences of CCDS tools - Surveys - 6 months | Provider surveys at 6 months post-CCDS implementation
  Provider survey questions will explore any unintended consequences of the CCDS tools. There is no published specific tool or scale that will be used.
Unintended consequences of CCDS tools - Surveys - 12 months | Provider surveys at 12 months post-CCDS implementation
  Provider survey questions will explore any unintended consequences of the CCDS tools. There is no published specific tool or scale that will be used.
Unintended consequences of CCDS tools - Interviews 6 months | Provider surveys and interviews at 6 months post-CCDS implementation
  Provider interview questions will explore any unintended consequences of the CCDS tools. There is no specific tool or scale that will be used.
Unintended consequences of CCDS tools - Interviews 12 months | Provider surveys and interviews at 12months post-CCDS implementation
  Provider interview questions will explore any unintended consequences of the CCDS tools. There is no specific tool or scale that will be used.
Impact of CCDS tools on quality of care - Surveys - 6 months | Provider surveys at 6 months post-CCDS implementation
  Provider survey questions will explore provider's subjective assessment of impact of the CCDS tools on the quality of care. There is no specific tool or scale that will be used.
Impact of CCDS tools on quality of care - Surveys - 12 months | Provider surveys at 12 months post-CCDS implementation
  Provider survey questions will explore provider's subjective assessment of impact of the CCDS tools on the quality of care. There is no specific tool or scale that will be used.
Impact of CCDS tools on quality of care - Interviews - 6 months | Provider interviews at 6 months post-CCDS implementation
  Provider interview questions will explore provider's subjective assessment of impact of the CCDS tools on the quality of care. There is no specific tool or scale that will be used.
Impact of CCDS tools on quality of care - Interviews - 12 months | Provider interviews at 12 months post-CCDS implementation
  Provider interview questions will explore provider's subjective assessment of impact of the CCDS tools on the quality of care. There is no specific tool or scale that will be used.
Adoption of CCDS tools | Provider surveys post-CCDS implementation
  Provider survey questions will address if providers reference the guidelines, if providers have encountered the CCDS alerts, the frequency with which they encounter the CCDS alerts, resources used to learn about the guidelines, and willingness and comfort using the CCDS alert recommendations. There is no specific score or scale being used for this outcome.
Barriers to CCDS implementation - Surveys - 6 months | Provider surveys and interviews at 6 months post-CCDS implementation
  Surveys will explore barriers to CCDS implementation at the individual, unit, and hospital levels.
Barriers to CCDS implementation - Surveys - 12 months | Provider surveys and interviews at 12 months post-CCDS implementation
  Surveys will explore barriers to CCDS implementation at the individual, unit, and hospital levels.
Barriers to CCDS implementation - Interviews - 6 months | Provider interviews at 6 months post-CCDS implementation
  Interviews will explore barriers to CCDS implementation at the individual, unit, and hospital levels. Provider interviews will also inquire about enabling factors in the following areas: CCDS tool delivery and intended use, time and resources needed to integrate the CCDS tools.
Barriers to CCDS implementation - Interviews - 12 months | Provider interviews at 12 months post-CCDS implementation
  Interviews will explore barriers to CCDS implementation at the individual, unit, and hospital levels. Provider interviews will also inquire about enabling factors in the following areas: CCDS tool delivery and intended use, time and resources needed to integrate the CCDS tools.
Enabling factors to CCDS implementation - Surveys - 6 months | Provider surveys at 6 months post-CCDS implementation
  Surveys will explore enabling factors to CCDS implementation at the individual, unit, and hospital levels.
Enabling factors to CCDS implementation - Surveys - 12 months | Provider surveys at 12 months post-CCDS implementation
  Surveys will explore enabling factors to CCDS implementation at the individual, unit, and hospital levels.
Enabling factors to CCDS implementation - Interviews - 6 months | Provider interviews at 6 months post-CCDS implementation
  Interviews will explore enabling factors to CCDS implementation at the individual, unit, and hospital levels. Provider interviews will inquire about enabling factors in the following areas: CCDS tool delivery and intended use, time and resources needed to integrate the CCDS tools.
Enabling factors to CCDS implementation - Interviews - 12 months | Provider interviews at 12 months post-CCDS implementation
  Interviews will explore enabling factors to CCDS implementation at the individual, unit, and hospital levels. Provider interviews will inquire about enabling factors in the following areas: CCDS tool delivery and intended use, time and resources needed to integrate the CCDS tools.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Lucile Packard Children's Hospital, Stanford University, Palo Alto, California
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Because PEDSnet is not a public data repository, individual-level datasets are not typically released publicly outside of the network. Due to the complexity and privacy concerns associated with electronic health record data, certified PEDSnet data scientists lead the execution of all data analyses. While the data generated for this study cannot be shared publicly, our study team will make every effort to assist interested investigators and teams in leveraging the PEDSnet network to collaborate to obtain the entire dataset from this study or subset of data necessary for conducting secondary analyses or in answering a new, intended study question. Our study team will provide a final report(s) on our research findings and the investigators will relate that data can be made available for subsequent analyses through PEDSnet and provide necessary contact information to submit a Collaboration Request through PEDSnet or Dr. Steffen.

DOCUMENTS (4):
  • Informed Consent Form: Informed consent form: post implementation survey (2024-05-30): https://cdn.clinicaltrials.gov/large-docs/74/NCT07108374/ICF_000.pdf
  • Informed Consent Form: Informed Consent Form: post implementation interview (2024-05-30): https://cdn.clinicaltrials.gov/large-docs/74/NCT07108374/ICF_001.pdf
  • Informed Consent Form: Pre-Implementation Survey (2024-11-26): https://cdn.clinicaltrials.gov/large-docs/74/NCT07108374/ICF_002.pdf
  • Informed Consent Form: Informed Consent Form: Practice Impact Survey (2024-11-26): https://cdn.clinicaltrials.gov/large-docs/74/NCT07108374/ICF_003.pdf